CLINICAL TRIAL: NCT02786173
Title: Peripheral Registry of Endovascular Clinical Outcomes
Brief Title: Peripheral Registry of Endovascular Clinical Outcomes "The PRIME Registry"
Acronym: PRIME
Status: Completed | Type: Observational
Sponsor: Metro Health, Michigan (Other)
Collaborators: C. R. Bard (Industry); Abbott Medical Devices (Industry); Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: PRIME
Record Dates: First submitted 2016-05-17; First posted 2016-05-30 (Estimated); Last update posted 2023-03-13 (Actual); Status verified 2022-03

CONDITIONS: Peripheral Arterial Disease; Peripheral Vascular Disease; Critical Limb Ischemia
Keywords: PRIME; PAD; PVD; Observational; CLI; PRIME Registry
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases; Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The PRIME Registry is a multi-center, observational study designed to evaluate immediate and long-term outcomes (36 months) of endovascular revascularization in patients with critical limb ischemia (CLI) and advanced peripheral artery disease (PAD).

DETAILED DESCRIPTION:
The Peripheral RegIstry of Endovascular Clinical OutcoMEs (PRIME Registry) represents the collaborative effort among seven centers across the US with the goal of reaching 10 sites globally. PRIME explores all aspects of advanced peripheral arterial disease (PAD) and critical limb ischemia (CLI) care including the collection of comprehensive clinical, diagnostic, procedural, and follow-up data for three years following an index endovascular procedure. Data collection activities began in January of 2013 with the goal of collecting data on 1500 subjects. Analysis of this multi-site registry will produce generalizable findings that describe the clinical epidemiology and management practices of advanced PAD and CLI patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are to receive or have received lower extremity endovascular intervention
* Rutherford III-VI Classification
* Ability to provide informed consent within 30 day prior to 60 days post index endovascular intervention.
* Ability to follow up at enrollment site.

Exclusion Criteria:

* Inability or unwillingness to consent for participation in the registry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are to receive or have received lower extremity endovascular treatment for peripheral artery disease.
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Amputation free survival rates | At 36 month follow-up visit

SECONDARY OUTCOMES:
Access site and procedural complications | At 36 month follow-up visit
Target lesion revascularization | At 36 month follow-up visit
Target vessel revascularization | At 36 month follow-up visit
Procedural success | At 36 month follow-up visit

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Orlando Health, Orlando, Florida
  - Prairie Heart, Springfield, Illinois
  - Metro Health Hospital, Wyoming, Michigan
  - Cox Health, Springfield, Missouri
  - Rex Healthcare, Raleigh, North Carolina
  - The Hospitals of Providence, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT02786173/Prot_SAP_001.pdf